CLINICAL TRIAL: NCT04694651
Title: A National Survey of Potential Acceptance of COVID-19 Vaccines in Healthcare Workers in Egypt
Brief Title: Potential Acceptance of COVID-19 Vaccines in Healthcare Workers in Egypt
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aliae AR Mohamed Hussein, Professor of Pulmonology, Assiut University
Other Study IDs: AssiutU18
Record Dates: First submitted 2020-12-20; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Covid19
Keywords: COVID-19; Healthcare workers; COVID-19 vaccines; Vaccine; Acceptance
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The COVID-19 pandemic is expected to remain as a public health threat and economic burden all over the world. The available proposed vaccines are still lacking large randomized controlled trials testing its efficacy and safety. Thus, the acceptance of vaccination between citizens as well as healthcare workers is not guaranteed. As the vaccine is starting to be distributed the acceptance of healthcare givers should be measured as they are usually the front line facing the problem and they have a responsibility to explain the need of immunization to the rest of population.

Strategies to enhance the acceptance and trust of the available vaccines may be needed.

ELIGIBILITY:
Inclusion Criteria: Healthcare workers

-

Exclusion Criteria:

* None healthcare workers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants were recruited by Consensus Strategies through online survey to avoid coverage bias.
  Doctors, nurses, laboratory workers and radiology technicians were included
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-01-30 (Estimated); Study Completion 2021-02-15 (Estimated)

PRIMARY OUTCOMES:
Measure frequency of acceptance of vaccination | 6 months
  number of healthcare worker agreeing to take the vaccine

SECONDARY OUTCOMES:
Describe causes of refusal of vaccination | 6 months
  answer a questionnaire of the causes of avoidance of vaccine

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - AssiutU, Asyut
  - Aliae AR Mohamed-Hussein, Asyut